CLINICAL TRIAL: NCT04353804
Title: Returning to Everyday Tasks Utilizing Rehabilitation Networks-III Pilot Randomized Clinical Trial (RETURN-III Pilot RCT)
Brief Title: Returning to Everyday Tasks Utilizing Rehabilitation Networks-III (RETURN-III)
Acronym: RETURN-III
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2992-R; 1506673-1 (Other: TVHS IRB); I01RX002992-01A2 (NIH); 230960 (Other: VUMC IRB)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Rehabilitation; ICU Survivorship; Intensive Care Unit; ICU
Keywords: Cognitive Rehabilitation; ICU Survivorship; Intensive Care Unit; ICU

STUDY DESIGN:
Intervention Model Description: The RETURN-III study will randomize medical and surgical VA ICU survivors to either 12-weeks of intervention using Computerized Cognitive Rehabilitation (CCR), or control of non-specific computer games.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The result of this randomization will be double-blinded, both to the study personnel and participants. All participants will access the computerized cognitive rehabilitation software (or control programs) via the same mechanism. Only specific support staff provided by our industry partner for purposes of training participants on the devices will have knowledge of the participant's randomization category other than the biostatisticians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computerized Cognitive Rehabilitation (Experimental): Computerized Cognitive Rehabilitation
  Interventions: Other: Treatment Arm: Computerized Cognitive Rehabilitation
- Active Control computer games (Active Comparator): Active Control computer games
  Interventions: Other: Active Control computer games

INTERVENTIONS:
Other: Treatment Arm: Computerized Cognitive Rehabilitation — Treatment Arm: Computerized Cognitive Rehabilitation
  Arms: Computerized Cognitive Rehabilitation
Other: Active Control computer games — Active Control computer games
  Arms: Active Control computer games

SUMMARY:
Millions of patients survive care in medical and surgical Intensive Care Units (ICUs) every year, only to suffer from a new or accelerated dementia-like process, called post-ICU long-term cognitive impairment (ICU-LTCI). ICU-LTCI causes considerable problems with personal relationships, return to work, and everyday tasks, such as managing medicines and money. No treatment for these patients is currently available. Technology using computerized cognitive rehabilitation could improve ICU-LTCI by harnessing the healing potential of the brain (i.e., neuroplasticity). This intervention is scalable, portable, and economical. The investigators will evaluate the effectiveness of computerized cognitive rehabilitation in a randomized controlled trial of 160 VA patients with ICU-LTCI. The investigators hypothesize that this intervention could improve cognition, and brain structure shown by MRI. This research has high potential to influence rehabilitation strategies for Veteran and civilian ICU survivors.

DETAILED DESCRIPTION:
Over a lifetime, an average American will be admitted to an intensive care unit (ICU) twice, will spend nearly a week in an ICU during their last six months of life, and will have a one in five chance of an ICU-related death. Of those millions who annually survive critical illness, ICU survivorship is marked by an inability to manage medication, handle finances, live independently, and maintain employment due to post-ICU long-term cognitive impairment (ICU-LTCI).

Data from the investigators' group and others show that 50% of ICU survivors suffer from ICU-LTCI. The investigators' Veterans Affairs (VA) Merit Award funded research, "Measuring the Incidence and determining risk factors for Neuropsychological Dysfunction in ICU Survivors" (MIND-ICU) study, helped define the epidemiology of this persistent and progressive chronic brain dysfunction that affects both executive function and memory domains of cognition. Among survivors from medical and surgical ICUs, 40% have impairments rivaling moderate traumatic brain injury, and 30% have impairments similar to mild-moderate Alzheimer's disease. The MIND-ICU study indicates that the number of Veterans who develop ICU-LTCI is as high as the number of new traumatic brain injury diagnoses among all Active Duty, National Guard, and Reserves of the Army, Navy, Air Force and Marine Corps. For a public health problem of this magnitude, there is a driving unmet need to find solutions for ICU-LTCI.

The investigators' pilot randomized "Returning to Everyday Tasks Utilizing Rehabilitation Networks-I" (RETURN-I) Study showed that a 12-week cognitive rehabilitation intervention (vs. controls) improved executive dysfunction. Next, the investigators transformed this non-computerized, resource-intensive strategy into a novel, efficient, and scalable Computerized Cognitive Rehabilitation (CCR) method. This plasticity-based adaptive CCR was applied to a case-series of ICU survivors which signaled improvements across multiple cognitive domains.

Building on nearly two decades of aging brain research with the VA-Tennessee Valley Geriatric Research, Education and Clinical Center (GRECC), the investigators now propose a Phase II randomized controlled trial (RCT) to investigate the efficacy of CCR for survivors with ICU-LTCI. The Returning to Everyday Tasks Utilizing Rehabilitation Networks-III Study (RETURN-III Study) will be the next logical data-driven approach to develop and offer innovative real-world solutions for civilians and Veterans surviving critical illness with disabling ICU-LTCI.

To test these hypotheses, the RETURN-III study will randomize medical and surgical VA ICU survivors to either intervention using CCR, or control of non-specific computer games. At three, and twelve months post-randomization, trained research personnel blinded to group assignment will use a validated battery to assess global cognition [primary outcome].

ELIGIBILITY:
Inclusion Criteria:

* Adults with a recent ICU stay (Medical or Surgical) requiring treatment for respiratory failure and/or shock (i.e., high-risk population)
* No longer requiring ICU-level care

Exclusion Criteria:

* No history of pre-existing severe cognitive impairment (IQCODE<3.3, documentation in medical record)
* Unwilling to commit to participation in the intervention
* Under consideration for hospice
* Primary residence over 100 miles from enrolling site if the patient is unwilling to return to the enrolling site for follow-up
* Homeless without a secondary contact available
* Severe substance abuse or neuropsychiatric disorder of a severity that prevents independent living
* Active suicidal ideation
* Any past or present behavior that may be deemed a safety risk for follow-up
* Blind, deaf, or unable to understand/communicate in English
* Required ICU level care less than 24 hours
* Not capable of completing computer-based training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Global Cognitive Composite Score | 3 months
  Global Cognitive Composite Score derived from the composite score provided by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS, range 40-160). The higher the number, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: E. Wesley Ely, MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN; Mayur B Patel, MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (2):
- United States (2):
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share data de-identified after study publication in accordance to clinical trial best practices and complying with federal guidelines for research.
Supporting Information: Study Protocol, SAP
Time Frame: We will share data de-identified >12 months after study publication in accordance to clinical trial best practices and complying with federal guidelines for research.
Access Criteria: We will share data de-identified after study publication in accordance to clinical trial best practices and complying with federal guidelines for research for an unlimited period of time.